CLINICAL TRIAL: NCT02744794
Title: Evaluation of a New Dermal Cryotherapy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R2 Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-15-001
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Skin Lightening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Treatment with cryotherapy (Experimental): Treatment with dermal cooling system.
  Interventions: Device: Dermal Cooling System

INTERVENTIONS:
Device: Dermal Cooling System — Treatment with cryotherapy.

SUMMARY:
A pilot study to evaluate the feasibility of altering skin pigmentation using the Dermal Cooling System.

DETAILED DESCRIPTION:
This non-significant risk study is being performed to test the hypothesis that a new treatment concept, controlled localized cooling of the epidermal layer, can be used to lighten areas of the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject is willing to have up to 40 test sites treated on aesthetically discreet skin.
3. Subject is willing to use photoprotection (e.g., sun avoidance) of the treated areas during the duration of the follow-up period.
4. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Fitzpatrick skin type VI.
2. Physician prescribed, medical or surgical treatment in the area of intended treatment in the previous 6 months (e.g., hydroquinone, corticosteroids, laser surgery)
3. Artificial tanning in the area of intended treatment within 1 month (e.g., spray, lotion, tanning bed) or intention to use artificial tanning within the follow-up period
4. Dermatological conditions or scars in the location of the treatment sites
5. History of melanoma, personal or first degree relative
6. Known history of illness or adverse reaction to cold insult (e.g., cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria, Reynaud's disease.
7. History of abnormal wound healing or abnormal scarring
8. Inability or unwillingness to comply with study requirments.
9. Current enrollment in a clinical study of any other unapproved investigational drug or device.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Skin pigmentation changes | 90 days
  Changes in pigmentation graded using a 7-point standardized scale

SECONDARY OUTCOMES:
Evaluation of device- or procedure-related adverse events | 0 to 12 months
  Side effects, discomfort assessments both during treatment and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Tatsutani, PhD, Study Director — R2 Dermatology, Inc.
Locations (3):
- United States (3):
  - Center of Dermatology and Laser Surgery, Sacramento, California
  - Diablo Clinical Research, Walnut Creek, California
  - Bowes Dermatology, Miami, Florida

IPD SHARING:
Plan to Share IPD: No